CLINICAL TRIAL: NCT04179890
Title: UpSwinG: Real World Study on TKI Activity in Uncommon Mutations and Sequencing Giotrif®
Brief Title: The Study Observes How Long Patients With Non-small Cell Lung Cancer (NSCLC) Benefit From Treatment With Epidermal Growth Factor Tyrosine Kinase Inhibitor (EGFR-TKI) When Given Either for Uncommon Mutations or for Common Mutations in the Sequence Afatinib Followed by Osimertinib
Acronym: UpSwinG
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1200-0316
Record Dates: First submitted 2019-11-26; First posted 2019-11-27 (Actual); Results first posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2022-07

CONDITIONS: Non-squamous, Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Afatinib; Erlotinib Hydrochloride; Gefitinib; osimertinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Uncommon EGFR mutation cohort: This arm included patients with Non-Small Cell Lung Cancer (NSCLC) carrying uncommon mutations in the epidermal growth factor receptor (EGFR) who were treated with the following Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitors (EGFR-TKIs) as first or second-line therapy:
  * Afatinib (Gi(l)otrif®):50mg or 40mg or 30mg or 20mg tablet once daily as indicated in the approved labels of afatinib (Gi(l)otrif®).
  * Erlotinib (Tarceva®): 25mg or 100mg or 150mg tablet once daily as indicated in the approved labels of erlotinib (Tarceva®).
  * Gefitinib (IRESSA®): 250mg tablet once daily as indicated in the approved labels of gefitinib (IRESSA®).
  * Osimertinib (Tagrisso®): 80 mg or 40 mg tablets once daily as indicated in the approved labels of osimertinib).
  In the first- or second-line with a threshold of start of treatment of at least 12 months respectively prior to data entry.
  Interventions: Drug: Afatinib (Gi(l)otrif®); Drug: Erlotinib (Tarceva®); Drug: Gefitinib (IRESSA®); Drug: Osimertinib (Tagrisso®)
- Sequencing cohort: This arm included Non-Small Cell Lung Cancer (NSCLC) patients with epidermal growth factor receptor (EGFR) mutation positive who received the following treatment sequence:
  - Afatinib (Gi(l)otrif®): 50mg or 40mg or 30mg or 20mg tablet once daily as indicated in the approved labels of afatinib (Gi(l)otrif®) as first line therapy, in the case the T790M resistance mutation was developed (second line therapy) the patients received osimertinib (Tagrisso®): 80 mg or 40 mg tablets once daily as indicated in the approved labels of osimertinib; the threshold of start of osimertinib at least 10 months prior to data entry.
  Interventions: Drug: Afatinib (Gi(l)otrif®); Drug: Osimertinib (Tagrisso®)

INTERVENTIONS:
Drug: Afatinib (Gi(l)otrif®) — Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor (EGFR-TKI) as first or second-line therapy.
  Groups: Uncommon EGFR mutation cohort
Drug: Erlotinib (Tarceva®) — Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor (EGFR-TKI) as first or second-line therapy.
  Groups: Uncommon EGFR mutation cohort
Drug: Gefitinib (IRESSA®) — Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor (EGFR-TKI) as first or second-line therapy.
  Groups: Uncommon EGFR mutation cohort
Drug: Osimertinib (Tagrisso®) — Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor (EGFR-TKI) as first or second-line therapy.
  Groups: Uncommon EGFR mutation cohort
Drug: Afatinib (Gi(l)otrif®) — As first line therapy.
  Groups: Sequencing cohort
Drug: Osimertinib (Tagrisso®) — In the case the T790M resistance mutation was developed (second line therapy).
  Groups: Sequencing cohort

SUMMARY:
Non-interventional, multi-country, multi-centre cohort study based on existing data from medical records (paper or electronic) or electronic health records of patients with advanced NSCLC harbouring EGFR mutations and treated with an EGFR-TKI

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients
2. Diagnosed with Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor (EGFRTKI) naive advanced EGFR mutated non-small cell lung cancer (NSCLC),
3. treated for Epidermal Growth Factor Receptor (EGFR) mutated NSCLC within regular clinical practice.
4. Informed and privacy consent signature must be obtained depending on local regulations.

   More specific inclusion criteria for each cohort are the following:

   Uncommon mutation cohort:
5. Patients harbouring uncommon or compound EGFR mutations
6. Patients who started with either afatinib (Gi(l)otrif®), gefitinib (Iressa®), erlotinib (Tarceva®), or osimertinib (Tagrisso®) in the first- or second-line setting within regular clinical practice
7. Patients must have started EGFR-TKI treatment at least 12 months prior to data entry.

Sequencing cohort:

5. Patients with common EGFR mutations (Del19, L858R) 6. Patients were treated with afatinib (Gi(l)otrif®) in the first-line setting and for acquired T790M mutation with osimertinib in the second line; 7. Patients must have started osimertinib treatment at least 10 months prior to data entry.

Patients treated with osimertinib within an early access program/ compassionate use program (EAP/CUP) are allowed

Exclusion Criteria:

1. Patients treated for EGFR mutated NSCLC within a clinical trial or participated in GioTag study.
2. Patients with active brain metastases at start of EGFR-TKI therapy (independent of treatment line)
3. For uncommon mutation cohort: Patients treated with osimertinib with no further uncommon mutation than acquired T790M Further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients diagnosed with Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor (EGFRTKI) naïve advanced EGFR mutated non-small cell lung cancer (NSCLC),
Sampling Method: Non-Probability Sample
Enrollment: 462 (Actual)
Dates: Start 2019-12-17 (Actual); Primary Completion 2021-07-22 (Actual); Study Completion 2021-07-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Marsden Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents. Exceptions might apply, e.g. studies in products where Boehringer Ingelheim is not the license holder; studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials; studies conducted in a single center or targeting rare diseases (in case of low number of patients and therefore limitations with anonymization).
  For more details refer to: https://www.mystudywindow.com/msw/datatransparency

REFERENCES:
- [Derived] Popat S, Hsia TC, Hung JY, Jung HA, Shih JY, Park CK, Lee SH, Okamoto T, Ahn HK, Lee YC, Sato Y, Lee SS, Mascaux C, Daoud H, Marten A, Miura S. Tyrosine Kinase Inhibitor Activity in Patients with NSCLC Harboring Uncommon EGFR Mutations: A Retrospective International Cohort Study (UpSwinG). Oncologist. 2022 Apr 5;27(4):255-265. doi: 10.1093/oncolo/oyac022. PMID 35274704
- See also: Related Info — http://www.mystudywindow.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A Real world, non-interventional study based on existing data from medical records or electronic health records. The study aimed to collect more information on the benefit of individual Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitors (EGFR-TKIs) treatment for the uncommon mutations and the overall benefit for the sequential EGFR TKI treatment with afatinib and osimertinib for the common EGFR mutations on patients with Non-Small Cell Lung Cancer (NSCLC).
Pre-assignment Details: Every patient who fulfilled inclusion and exclusion criteria and agreed to participate in the study was selected until the required sample size was achieved. Deceased and untraceable patients were enrolled whenever possible and discussed with the local authorities.
Period: Overall Study
Arm/Group | Uncommon EGFR Mutation Cohort | Sequencing Cohort
Started (Reporting Enrolled Patients) | 255 | 207
Eligible Patients | 246 | 191
Completed | 246 | 191
Not Completed | 9 | 16
Not completed — Patients not harbouring uncommon or compound EGFR mutations | 3 | 0
Not completed — Patients who did not start EGFR-TKI treatment at least 12 months prior to data entry | 1 | 0
Not completed — Patients treated for EGFR mutated NSCLC within a clinical trial | 3 | 0
Not completed — Patients with active brain metastases at start of EGFR-TKI therapy | 2 | 0
Not completed — Patients not treated with afatinib in first-line or with osimertinib in second line | 0 | 8
Not completed — Patients not starting osimertinib treatment at least 10 months prior to data entry | 0 | 4
Not completed — Patients with active brain metastases at start of EGFR-TKI therapy (independent of treatment line) | 0 | 2
Not completed — Patients without common EGFR mutations (Del19, L858R) | 0 | 1
Not completed — Patients treated for EGFR mutated NSCLC within a clinical trial or participated in GioTag study | 0 | 1

BASELINE CHARACTERISTICS:
Population: Eligible Patients set (Uncommon mutation and common mutation cohorts): All enrolled patients meeting all the inclusion and exclusion criteria to be evaluable.
Groups:
- Total: Total of all reporting groups
Arm/Group | Uncommon EGFR Mutation Cohort | Sequencing Cohort | Total
Number analyzed (Participants) | 246 | 191 | 437
Age, Continuous [Mean (Standard Deviation); unit: Years] | 67.6 (11.0) | 61.4 (11.7) | 64.89 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 138 | 106 | 244
  Male | 108 | 85 | 193
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 206 | 118 | 324
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 23 | 55 | 78
  More than one race | 0 | 2 | 2
  Unknown or Not Reported | 17 | 15 | 32

OUTCOME MEASURES:

1. Primary Outcome: Time on Treatment With Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitor (EGFR-TKI)
Description: Uncommon Mutation Cohort: Time on treatment with EGFR-TKI assessed as the time from start of EGFR-TKI treatment until the end of treatment or death by any cause is reported.
  Common mutation cohort: Time on treatment with EGFR-TKI assessed as the time from start of afatinib (Gi(l)otrif®) as first-line treatment until the end of the second line treatment (the last dose of osimertinib) or death date by any cause.
  Time on treatment was analysed using Kaplan-Meier method, and the median was tabulated along with two-sided 95% confidence interval using the Greenwood's variance estimate.
Time Frame: Up to 13 years for Uncommon EGFR mutation cohort and up to 6 years for the Sequencing Cohort.
Population: Eligible Patients set (Uncommon mutation cohort): All enrolled patients meeting all the inclusion and exclusion criteria to be evaluable.
  Eligible Patients set (Sequencing cohort): All enrolled patients meeting all the inclusion and exclusion criteria to be evaluable.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Uncommon EGFR Mutation Cohort | Sequencing Cohort
Number analyzed (Participants) | 246 | 191
Months | 9.89 [7.75 to 11.56] | 27.7 [23.95 to 30.23]

2. Secondary Outcome: Uncommon Epidermal Growth Factor Receptor (EGFR) Mutation Cohort: Overall Response Rate to Index Line Treatment
Description: Overall response rate (ORR) using RECIST criteria as assessed by investigator. ORR to index line Epidermal Growth Factor Receptor-Tyrosine Kinase Inhibitor (EGFR-TKI) treatment is reported (ORR is defined as number of patients with complete or partial response evaluated by Response Evaluation Criteria In Solid Tumors Criteria (RECIST 1.1)).
  (Per RECIST 1.1: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR).
Time Frame: Up to 13 years.
Population: Eligible Patients set (Uncommon mutation cohort): All enrolled patients meeting all the inclusion and exclusion criteria to be evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Uncommon EGFR Mutation Cohort
Number analyzed (Participants) | 246
Participants | 96

3. Secondary Outcome: Sequencing Cohort: Overall Response Rate to First Line Afatinib
Description: Overall response rate (ORR) using RECIST criteria as assessed by investigator. Overall response rate to first line afatinib treatment for the Common Epidermal Growth Factor Receptor (EGFR) mutation cohort is reported. (ORR is defined as number of patients with complete or partial response evaluated by Response Evaluation Criteria In Solid Tumors Criteria (RECIST 1.1)).
  (Per RECIST 1.1: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR).
Time Frame: Up to 6 years.
Population: Eligible Patients set (Sequencing cohort): All enrolled patients meeting all the inclusion and exclusion criteria to be evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Sequencing Cohort
Number analyzed (Participants) | 191
Participants | 131

4. Secondary Outcome: Sequencing Cohort: Overall Response Rate to Second-line Treatment Osimertinib
Description: Overall response rate (ORR) using RECIST criteria as assessed by investigator. Overall response rate to second-line treatment (Osimertinib) is reported. (ORR is defined as number of patients with complete or partial response evaluated by Response Evaluation Criteria In Solid Tumors Criteria (RECIST 1.1)).
  (Per RECIST 1.1: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR).
Time Frame: Up to 6 years.
Population: as for outcome 3
Measure: Count of Participants; unit: Participants
Arm/Group | Sequencing Cohort
Number analyzed (Participants) | 191
Participants | 75

5. Secondary Outcome: Overall Survival
Description: Uncommon Mutation Cohort: Overall survival since index line treatment start of Tyrosine Kinase Inhibitor (TKI) medication administered per generation until death date by any cause or the end of index line is reported. Sequencing cohort: Overall survival for since first-line afatinib treatment start until death date by any cause or the end of index line. Kaplan-Meier estimates of quartiles of time to death were computed (with their 95% Confidence Intervals, using Greenwood's variance estimate.
Time Frame: Up to 13 years for Uncommon EGFR mutation cohort and up to 6 years for the Sequencing Cohort.
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Uncommon EGFR Mutation Cohort | Sequencing Cohort
Number analyzed (Participants) | 246 | 191
Months | 24.44 [20.24 to 28.16] | 36.50 [32.85 to 41.76]

6. Secondary Outcome: Number of Participants for Each Type of Biological Samples Used for Mutation Detection at First Line Treatment Start
Description: Number of participants for each type of biological samples used for mutation detection at first line treatment start is reported.
  The reported types of biological samples are:
  * Tissue, histological sample (solid biopsy);
  * Cytological sample;
  * Blood (liquid biopsy);
  * Other and
  * Unknown.
Time Frame: At first-line treatment start (i.e. between 2007 and 2019 for the Uncommon Epidermal Growth Factor Receptor (EGFR) mutation cohort and between 2014 and 2018 for Sequencing Cohort).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Uncommon EGFR Mutation Cohort | Sequencing Cohort
Number analyzed (Participants) | 246 | 191
Participants
  Tissue, Histological sample (solid biopsy) | 212 | 160
  Cytological sample | 32 | 19
  Blood (liquid biopsy) | 3 | 6
  Other | 2 | 2
  Unknown | 3 | 6

7. Secondary Outcome: Number of Participants for Each Category of Methodology Used for Mutational Testing at First Line Treatment Start
Description: Number of participants for each type of methodologies used for mutational testing is reported.
  The reported types of methodology are:
  * Amplification Refractory Mutation System (ARMS);
  * Polymerase Chain reactions (PCR)-based techniques;
  * Sequencing;
  * Next-Generation Sequencing (NGS);
  * Other;
  * Unknown.
Time Frame: At first-line treatment start (i.e. between 2007 and 2019 for the Uncommon Epidermal Growth Factor Receptor (EGFR) mutation cohort and between 2014 and 2018 for the Sequencing Cohort).
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Uncommon EGFR Mutation Cohort | Sequencing Cohort
Number analyzed (Participants) | 246 | 191
Participants
  Amplification Refractory Mutation System (ARMS) | 4 | 4
  PCR-based techniques | 155 | 122
  Sequencing | 39 | 15
  Next-Generation Sequencing (NGS) | 20 | 8
  Unknown | 42 | 41
  Other | 0 | 1

8. Secondary Outcome: Uncommon Mutation Cohort: Time on Treatment Until Failure of Second-line (TTF2)
Description: Time on treatment until failure of second-line (TTF2), defined as time elapsed from start of first-line treatment (regardless the type of treatment) to stop of second-line (regardless of the type of treatment) or death by any cause is reported. Kaplan-Meier estimates of quartiles of time to second-line treatment failure were computed (with their 95% Confidence Intervals, using Greenwood's variance estimate).
Time Frame: From start of first-line treatment to stop of second-line or death by any cause, up to 13 years.
Population: Eligible Patients set (Uncommon mutation cohort): All enrolled patients meeting all the inclusion and exclusion criteria to be evaluable and who were initiated on a second line treatment.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Uncommon EGFR Mutation Cohort
Number analyzed (Participants) | 140
Months | 14.46 [13.24 to 18.00]

9. Secondary Outcome: Number of Participants for Each Type of Biological Samples Used for Mutation Detection at Second Line Treatment Start
Description: Number of participants for each type of biological samples used for mutation detection at second line treatment start is reported.
  The reported types of biological samples are:
  * Tissue, Histological sample (solid biopsy);
  * Cytological sample;
  * Blood (liquid biopsy);
  * Not applicable-Clinical evaluation;
  * Other;
  * Unknown. Not applicable - Clinical evaluation: The uncommon Epidermal Growth Factor Receptor (EGFR) mutational status had become available after Progression on conventional second-line therapy. Erlotinib was given as state of the art second-line therapy in 2014, and an EGFR mutation was clinically suspected due to the Long-Lasting response. However, due to the unavailability of tumor tissue, this could be proven only after liquid biopsy had subsequently become available at the center in 2016.
  For the Sequencing cohort second-line treatment start is initiated by the beginning of the therapy with Osimertinib.
Time Frame: At second-line treatment start (i.e. between 2007 and 16-Jul-2020 for "Uncommon EGFR mutation cohort" and between 2014 and 23-Oct-2020 for the "Sequencing Cohort
Population: Eligible Patients set: All enrolled patients meeting all the inclusion and exclusion criteria to be evaluable and who were initiated on a second line treatment. For the Uncommon EGFR mutation cohort only patients with >1 Non-Small Cell Lung Cancer (NSCLC) with re-evaluated mutational status.
Measure: Count of Participants; unit: Participants
Arm/Group | Uncommon EGFR Mutation Cohort | Sequencing Cohort
Number analyzed (Participants) | 34 | 191
Participants
  Tissue, Histological sample (solid biopsy) | 22 | 93
  Cytological sample | 3 | 18
  Blood (liquid biopsy) | 8 | 57
  Not applicable - Clinical evaluation | 1 | 0
  Other | 0 | 7
  Unknown | 0 | 19

10. Secondary Outcome: Number of Participants for Each Type of Biological Samples Used for Mutation Detection at Second Line Treatment Stop/End of Observation
Description: Number of participants for each type of biological samples used for mutation detection at second line treatment stop/end of observation is reported.
  The reported categories of biological samples are:
  * Tissue, Histological sample (solid biopsy);
  * Cytological sample;
  * Blood (liquid biopsy);
  * Other.
Time Frame: At second-line treatment start (i.e. between 2007 and 16-Jul-2020 for Uncommon Epidermal Growth Factor Receptor (EGFR) mutation cohort and between 2014 and 23-Oct-2020 for the Sequencing Cohort).
Population: Eligible Patients set: All enrolled patients meeting all the inclusion and exclusion criteria to be evaluable. For the Uncommon EGFR mutation cohort eligible patients with >1 Non-Small Cell Lung Cancer (NSCLC) line with re-evaluated mutational status are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Uncommon EGFR Mutation Cohort | Sequencing Cohort
Number analyzed (Participants) | 10 | 191
Participants
  Tissue, Histological sample (solid biopsy) | 5 | 9
  Blood (liquid biopsy) | 4 | 9
  Other | 1 | 0
  Cytological sample | 0 | 1

11. Secondary Outcome: Uncommon Cohort: Number of Participants for Each Type of Biological Samples Used for Mutation Detection at Index Therapy Start
Description: Number of participants for each type of biological samples used for mutation detection at index therapy start (index therapy refers to therapy switch from first-line chemotherapy to second-line Epidermal Growth Factor Receptor-Tyrosine Kinase Inhibitor (EGFR-TKI) therapy (index line)) is reported.
  The reported categories of biological samples are:
  * Tissue, Histological sample (solid biopsy);
  * Cytological sample;
  * Blood (liquid biopsy);
  * Other and
  * Unknown.
Time Frame: Up to 13 years.
Population: Eligible Patients set: All enrolled patients meeting all the inclusion and exclusion criteria to be evaluable. 16 patients in the Uncommon EGFR mutation cohort who switched from first-line chemotherapy to second-line EGFR-TKI therapy for which EGFR mutational status was not re-evaluated at start of second-line treatment were not included in this group.
Measure: Count of Participants; unit: Participants
Arm/Group | Uncommon EGFR Mutation Cohort
Number analyzed (Participants) | 230
Participants
  Tissue, Histological sample (solid biopsy) | 199
  Cytological sample | 29
  Blood (liquid biopsy) | 2
  Other | 2
  Unknown | 3

12. Secondary Outcome: Number of Participants for Each Type of Methodology Used for Mutational Testing at Second-line Treatment Start
Description: Number of participants for each type of methodology used for mutational testing at second-line treatment start is reported.
  The reported types of methodologies are:
  * Amplification Refractory Mutation System (ARMS);
  * Polymerase Chain Reaction (PCR)-based techniques;
  * Sequencing;
  * Next-Generation Sequencing (NGS);
  * Other;
  * Unknown/Not applicable- Clinical evaluation.
Time Frame: At second-line treatment start (i.e. between 2007 and 16-Jul-2020 for Uncommon Epidermal Growth Factor Receptor-Tyrosine Kinase Inhibitor (EGFR) mutation cohort and between 2014 and 23-Oct-2020 for the Sequencing Cohort).
Population: as for outcome 9
Measure: Count of Participants; unit: Participants
Arm/Group | Uncommon EGFR Mutation Cohort | Sequencing Cohort
Number analyzed (Participants) | 34 | 191
Participants
  PCR-based techniques | 23 | 121
  Sequencing | 2 | 2
  Next-Generation Sequencing (NGS) | 3 | 13
  Unknown/Not applicable- Clinical evaluation | 6 | 51
  Amplification Refractory Mutation System (ARMS) | 0 | 3
  Other | 0 | 1

13. Secondary Outcome: Number of Participants for Each Type of Methodology Used for Mutational Testing at Second-line Treatment Stop/End of Observation
Description: Number of participants for each type of methodology used for mutational testing is reported.
  The reported types of methodologies are:
  * Polymerase Chain Reaction (PCR)-based techniques;
  * Next-Generation Sequencing (NGS);
  * Unknown.
Time Frame: At second-line treatment stop/end of observation (i.e. between 2007 and 16-Jul-2020 for Uncommon Epidermal Growth Factor Receptor (EGFR) mutation cohort and between 2014 and 23-Oct-2020 for the Sequencing Cohort).
Population: Eligible Patients set: All enrolled patients meeting all the inclusion and exclusion criteria to be evaluable.
Measure: Count of Participants; unit: Participants
Arm/Group | Uncommon EGFR Mutation Cohort | Sequencing Cohort
Number analyzed (Participants) | 10 | 16
Participants
  PCR-based techniques | 7 | 11
  Next-Generation Sequencing (NGS) | 2 | 2
  Unknown | 1 | 3

14. Secondary Outcome: Uncommon Mutation Cohort: Number of Participants for Each Type of Methodology Used for Mutation Detection at Index Therapy Start
Description: Number of participants for each type of methodology used for mutation detection at index therapy start is reported. Index therapy refers to therapy switch from first-line chemotherapy to second-line Epidermal Growth Factor Receptor-Tyrosine Kinase Inhibitor (EGFR-TKI) therapy (index line).
  The reported categories of methodology are:
  * Amplification Refractory Mutation System (ARMS),
  * Polymerase chain reaction based techniques (PCR-based techniques),
  * Sequencing,
  * Next-Generation Sequencing (NGS),
  * Unknown.
Time Frame: Up to 13 years.
Population: Eligible Patients set: All enrolled patients meeting all the inclusion and exclusion criteria to be evaluable. 16 patients in the "Uncommon EGFR mutation cohort" who switched from first-line chemotherapy to second-line EGFR-TKI therapy for which EGFR mutational status was not re-evaluated at start of second-line treatment were not included in this group.
Measure: Count of Participants; unit: Participants
Arm/Group | Uncommon EGFR Mutation Cohort
Number analyzed (Participants) | 230
Participants
  Amplification Refractory Mutation System (ARMS) | 4
  PCR-based techniques | 146
  Sequencing | 34
  Next-Generation Sequencing (NGS) | 18
  Unknown | 41

15. Secondary Outcome: Uncommon Mutation Cohort: Number of Participants for Each Type of Methodology Used for Mutation Detection at Start of First-line Chemotherapy Before Index Line
Description: Number of participants for each type of methodology used for mutation detection at start of first-line chemotherapy before index line is reported.
  The reported types of methodologies are:
  * PCR-based techniques;
  * Sequencing;
  * Next-Generation Sequencing (NGS);
  * Unknown.
  Index therapy refers to therapy switch from first-line chemotherapy to second-line Epidermal Growth Factor Receptor-Tyrosine Kinase Inhibitor (EGFR-TKI) therapy (index line).
Time Frame: At start of first-line chemotherapy before index line (i.e. between 2007 and 2019).
Population: Eligible Patients set: All enrolled patients meeting all the inclusion and exclusion criteria to be evaluable. Only patients switching from first-line chemotherapy to second-line EGFR-TKI therapy (index line) for which EGFR mutational status was not re-evaluated at start of second-line treatment are reported.
Measure: Count of Participants; unit: Participants
Arm/Group | Uncommon EGFR Mutation Cohort
Number analyzed (Participants) | 16
Participants
  PCR-based techniques | 9
  Sequencing | 5
  Next-Generation Sequencing (NGS) | 2
  Unknown | 1

16. Secondary Outcome: Uncommon Mutation Cohort: Number of Participants for Each Type of Biological Samples Used for Mutation Detection at Start of First-line Chemotherapy Before Index Line
Description: Number of participants for each type of biological samples used for mutation detection at start of first-line chemotherapy before index line is reported. Index therapy refers to therapy switch from first-line chemotherapy to second-line Epidermal Growth Factor Receptor-Tyrosine Kinase Inhibitor (EGFR-TKI) therapy (index line).
  The reported types of biological samples are:
  * Tissue, Histological sample (solid biopsy);
  * Cytological sample, Blood (liquid biopsy).
Time Frame: At start of first-line chemotherapy before index line (i.e. between 2007 and 2019).
Population: as for outcome 15
Measure: Count of Participants; unit: Participants
Arm/Group | Uncommon EGFR Mutation Cohort
Number analyzed (Participants) | 16
Participants
  Tissue, Histological sample (solid biopsy) | 13
  Cytological sample | 3
  Blood (liquid biopsy) | 1

ADVERSE EVENTS:
Time Frame: From the start of the first-line treatment between 2007 and 2019, until Database Lock in 2021. Up to 14 years.
Description: A Safety analysis was included, reporting adverse drug reaction (ADR) information that was provided by the Pharmacovigilance (PV) Department at Boehringer Ingelheim, which was linked to patient data. The safety analysis included no adverse events beyond ADR and fatal adverse events (AEs). The safety analysis as per statistical analysis plan is reported on the overall enrolled patients set for those subjects that have not missing safety data.
Arm/Group | Sequencing Cohort | Uncommon EGFR Mutation Cohort
All-Cause Mortality (participants affected / at risk) | 0/44 | 0/35
Serious Adverse Events (participants affected / at risk) | 12/44 | 6/35
Other Adverse Events (participants affected / at risk) | 41/44 | 30/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sequencing Cohort (N=44) | Uncommon EGFR Mutation Cohort (N=35)
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Disease progression (General disorders) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 10 | 3
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sequencing Cohort (N=44) | Uncommon EGFR Mutation Cohort (N=35)
Diarrhoea (Gastrointestinal disorders) | 34 | 24
Stomatitis (Gastrointestinal disorders) | 13 | 12
Paronychia (Infections and infestations) | 17 | 12
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 6 | 12
Dry skin (Skin and subcutaneous tissue disorders) | 4 | 2
Rash (Skin and subcutaneous tissue disorders) | 19 | 7
Nausea (Gastrointestinal disorders) | 3 | 0
Inflammation (General disorders) | 3 | 0
Mucosal inflammation (General disorders) | 3 | 0
Oedema peripheral (General disorders) | 0 | 3
Decreased appetite (Metabolism and nutrition disorders) | 1 | 2
Dermatitis (Skin and subcutaneous tissue disorders) | 3 | 1
Nail fold inflammation (Skin and subcutaneous tissue disorders) | 0 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 2

LIMITATIONS AND CAVEATS:
As in all studies based on secondary use of data, the risk of missing data shall be taken into consideration. Stratified analyses include no formal testing for statistical significance since such analyses have a descriptive exploratory purpose. In fact, no a priori hypotheses were defined. Patient's duration of observation was different for each subject without specific censoring rules by protocol, and there were no limitations on time periods for starting treatments by protocol.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2020-06-20): https://cdn.clinicaltrials.gov/large-docs/90/NCT04179890/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-11): https://cdn.clinicaltrials.gov/large-docs/90/NCT04179890/SAP_001.pdf